CLINICAL TRIAL: NCT01545739
Title: Master Study of the Evia/Entovis HF-T Pacemaker
Brief Title: Evia/Entovis HF-T Master Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 57
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Indication for Cardiac Resynchronization Therapy (CRT)
Keywords: Pacemaker therapy; Cardiac resynchronisation therapy (CRT)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT pacemaker implantation
  Interventions: Device: Evia/Entovis HF-T pacemaker for CRT therapy

INTERVENTIONS:
Device: Evia/Entovis HF-T pacemaker for CRT therapy — Implantation of CRT pacemaker and standard follow-ups at pre-hospital discharge, and after 1, 3 and 6 months

SUMMARY:
The Evia HF-T and the Entovis HF-T are triple-chamber pacemakers for cardiac resynchronisation therapy (CRT-P). The objective of this study is to prove the safety and efficacy of these pacemakers. In particular, the left ventricular (LV) capture control feature is evaluated, which automatically measures the LV pacing threshold and subsequently adjusts the pacing output.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for CRT therapy
* Legal capacity and ability to consent
* Signed patient informed consent

Exclusion Criteria:

* Contraindication for CRT therapy
* ICD indication
* Age < 18 years
* Pregnant or breast-feeding woman
* Cardiac surgery planned within the next 6 months
* Life expectancy of less than 6 months
* Participating in another clinical study of an investigational cardiac drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for CRT therapy
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety: Serious Adverse Device Effect (SADE) free rate | Until 3 month follow-up
  While the investigator is asked to record all adverse events throughout the study, only the number of SADEs possibly or securely related to a device deficiency will be the basis for the calculation of the SADE free rate: (1-number of SADE divided by number of patients)%.
Efficacy of the left ventricular capture control feature (focus on threshold measurements) | At pre-hospital discharge, 1 and 3 month follow-up
  Absolute difference between the triggered automatic and manual pacing threshold in the left ventricle is smaller than 0.3 Volt.

SECONDARY OUTCOMES:
Efficacy of the left ventricular capture control feature (focus on pulse amplitude adjustment) | 1 and 3 month follow-up
  Rate of appropriate adjustment of the left ventricular (LV) pulse amplitude by the LV capture control feature is greater than 90%.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary